

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Feasibility of dietary magnesium replacement for prevention of hypomagnesemia in ovarian cancer patients receiving carboplatin chemotherapy 2018-1172

| Study Chair: | Lorenzo Cohen |
|--------------------|-----------------------|
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

### STUDY SUMMARY

A common side of effect of carboplatin-containing chemotherapy is hypomagnesemia low blood levels of magnesium in the blood that may cause weakness, muscle cramps, and/or irregular heartbeat).

The goal of this research study is to learn if adding foods that naturally contain magnesium to the diet of ovarian cancer patients who are receiving carboplatin-containing chemotherapy can increase the levels of magnesium in the blood and help prevent hypomagnesemia.

# This is an investigational study.

Increasing the amount of foods you eat that contain magnesium may help raise your magnesium blood levels and prevent the risk of hypomagnesemia. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. You may not wish to take part in the study if you have food allergies that prevent you from following the diet.

You can read a list of potential side effects below in the Possible Risks section of this consent.

Your participation in the study will be over after you have completed 6 cycles of carboplatin-containing chemotherapy as part of your standard care.

There is no cost to take part in the study.

You may choose not to participate in this study. You can continue to be treated at MD Anderson.

#### 1. STUDY DETAILS

Up to 50 participants will be enrolled in this study. All will take part at MD Anderson.

If you agree to take part in this study, information from your medical record (such as your age and weight/height, your medical history, cancer stage, and if you have had a surgical resection) will be collected.

You will be asked to complete a study questionnaire either on the phone, electronically via REDCap, or by mail on paper. The questionnaire will have questions about the foods you eat and it will take about 30 minutes to complete.

You will then be given 2 handouts. One handout will list the types of foods and drinks that are high in magnesium and the amount of magnesium per serving. You need to consume at least 400mg of magnesium total from these foods every day. You will also be given a handout of different recipes that you can use to help you during this time.

You will be contacted by a registered dietitian or study staff 1 time every week either by phone or by video interviews (such as Skype). During these calls, you will be asked what you ate in the last 24 hours and which magnesium-rich foods you ate. Each call should last about 10-20 minutes.

If your primary physician thinks it is needed, you may still receive a standard magnesium supplement as part of your standard care. If this is given, your doctor will discuss how and when the supplement is given, including its risks. If you receive a magnesium supplement, that information will be collected as part of this study.

As part of your standard care, blood will be drawn for routine tests (which will include a check of how much magnesium is in your blood) while you receive chemotherapy. As part of your participation in this study, the results of those routine tests and magnesium levels will be collected from your medical record.

#### 2. POSSIBLE RISKS

Although every effort will be made to keep **study data** safe, there is a chance that your personal health information could be lost or stolen. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

**Questionnaires** may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaire, you are encouraged to contact your doctor or the study chair.

This study may involve unpredictable risks to the participants.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-2933 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

# **Additional Information**

4. You may ask the study chair (Dr. Lorenzo Cohen, at 713-745-4260) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB - a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.

- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.

#### **Future Research**

Your personal information is being collected as part of this study. This information, or data, may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

Before being shared for future research, every effort will be made to remove your identifying information from any data. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data are used for future research. If this research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.

# <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and

study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:

- Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
- The IRB and officials of MD Anderson
- Study monitors and auditors who verify the accuracy of the information
- Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

| I understand the information in this consent form. I have had a chance consent form for this study, or have had it read to me. I have had a cabout it, ask questions, and talk about it with others as needed. I give permission to enroll me on this study. By signing this consent form, I any of my legal rights. I will be given a signed copy of this consent d | hance to think<br>the study chair<br>am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| LEGALLY AUTHORIZED REPRESENTATIVE (LAR) The following signature line should only be filled out when the partic the capacity to legally consent to take part in the study and/or sign to or her own behalf. | • |
| SIGNATURE OF LAR | DATE |
| PRINTED NAME and RELATIONSHIP TO PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be performed 2018-1172. | under Protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for vulnerable adult participants. If witnessing a pediatric participant, leave this line blank and sign on the witness to assent page in | |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or representative, using language that is understandable and appropriate have fully informed this participant of the nature of this study and its pand risks and that the participant understood this explanation. | te. I believe that I |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |

| <u>TRANSLATOR</u> | | | |
|---|---|---|---|
| I have translated the above in subtractions) into (Na obtaining and providing conse | and<br>ame of Language) | l assisted the peo | ople |
| consent process for this partic | | , and responses | daming the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLA | TOR [ | DATE |
| ☐ Please check here if the translator was a member of the research team. (If checked, a witness, other than the translator, must sign the witness line below.) | | | |
| SIGNATURE OF WITNESS T<br>(OTHER THAN TRANSLATO<br>OR STUDY CHAIR) | | ION [ | DATE |

PRINTED NAME OF WITNESS TO THE VERBAL TRANSLATION